CLINICAL TRIAL: NCT01510418
Title: Socialization of Adult Men With Congenital Hemophilia A or B: A Study to Examine Socialization Measures, the Role of Spouse/Significant Other and Health Related Quality of Life
Brief Title: Socialization of Adult Men With Congenital Hemophilia A or B
Acronym: PWBCD
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Aric Parnes, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 10-343
Record Dates: First submitted 2011-10-03; First posted 2012-01-16 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia; Spouse; Significant Other; Quality of Life
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Person with congenital bleeding disorder: Adult men with congenital hemophilia A or B
- Spouse/Significant Other: Spouse/significant other of person with congenital bleeding disorder participating in this study.

SUMMARY:
The goal of this pilot study is to understand the socialization of adult men with hemophilia living in the United States and their quality of life in order to improve comprehensive care for persons with congenital bleeding disorders. Studies in Europe suggest that despite medical, surgical, and biotechnology advances in care for persons with the congenital bleeding disorders hemophilia A and B, men with hemophilia have earlier work disability and health-related lower quality of life than men of the same age who do not have hemophilia in the general population. Congenital bleeding disorders are known to have medical and psychosocial impact not only in school but also in other activities, e.g. participation in sports beginning at a young age. The psychosocial impact of living with a congenital bleeding disorder has been studied and described in childhood. The support relationships in childhood include parents and primary family of origin and these supports are generally considered in pediatric comprehensive care models. Support relationships in adulthood have not been well described or studied. The role of spouse and significant others (SSO) of PWCBD in health care is of interest for the delivery of adult comprehensive care as well as to understand their contribution to the health-related quality of life of PWCBD. Additionally, this study seeks to learn of the impact of congenital bleeding disorders for the SSO. The study uses self-reported medical and social information questionnaires, health-related quality of life surveys, and confidential interview. Results of this study may guide how comprehensive care and support are provided to adult persons with congenital bleeding disorders by hemophilia treatment programs. This study focuses on PWCBD with hemophilia A or B as a model for the experience of persons with other congenital bleeding disorders.

DETAILED DESCRIPTION:
There are two groups (cohorts) in this study. One group is adult men with congenital hemophilia A or B who qualify for the study. The other group is their spouse or significant other (SSO) who are voluntarily identified by the person with congenital bleeding disorder for recruitment into the study.

For the adult men with congenital hemophilia A or B, the study involves a minimum of 2 visits and includes screening, medical history and physical exam review, completing confidential questionnaires and interview.

Eligible men with congenital hemophilia A or B (person with congenital bleeding disorder, PWCBD) are given the option to permit the investigator to contact their spouse or significant other (SSO) for participation in the study. If PWCBD has an SSO, the SSO is not required to participate in the study.

Spouse/significant other(SSO)of men with congenital hemophilia A or B may enter the study only if they have been voluntarily identified by their partner (PWCBD) and their partner has opted to allow investigator to contact them. For the SSO who chooses to participate in the study, the study will involve a minimum of one visit and includes completing confidential questionnaires and interview.

All participation including questionnaires and interview information collected is confidential and protected by health privacy information laws and records are de-identified.

The study is sponsored by a grant from The National Hemophilia Foundation.

ELIGIBILITY:
Eligibility criteria for person with congenital bleeding disorder(PWCBD, men with congenital hemophilia):

* Known diagnosis of congenital hemophilia A or B with or without inhibitor (defined by a plasma factor VIII or factor IX level below lower limits of normal and medical history consistent with diagnosis).
* Male age 21 years or older
* Willing to indicate if they have a spouse or significant other.
* Able to read, write and participate in interview on site.

Exclusion Criteria for PWCBD:

* Other bleeding disorder besides congenital hemophilia A or B

Eligibility criteria for spouses/significant other (SSO) participants in the study:

* A person in a relationship for a minimum of 9 months with the PWCBD participating in the study.
* PWCBD partner must be participating in the study.
* Willing to participate in questionnaire and interview on site.

Exclusion criteria for SSO:

- Biologically related to PWCBD participant (that is, not a parent, sibling, child or other biologically-related caregiver).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are two study populations:
  PWCBD: Person with congenital bleeding disorders are adult men with congenital hemophilia A or B who receive care in Massachusetts or who reside in the New England area or elsewhere and are willing to travel to the study site may be eligible for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Health related quality of life, description of support and networks. | 2 years
  Standard health-related quality of life questionnaires and interview are used to obtain primary outcome measure about PWCBD.

SECONDARY OUTCOMES:
Quality of life and description of role of SSO in health care of their PWCBD partner | 2 years
  Standardized quality of life questionnaire, social-medical questionnaire and interview of SSO are used to obtain this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Aric Parnes, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States